CLINICAL TRIAL: NCT06284590
Title: A Phase 2, Three-arm, Randomized Study of the Efficacy of Intratumorally Administered L19IL2 or L19TNF or L19IL2/L19TNF, All in Combination with Systemic Anti-PD1 Pembrolizumab, in Stage III and IV Unresectable Melanoma Patients with Resistance to or Progressing Upon Anti-PD1 Checkpoint Inhibitors and with Presence of Injectable Metastases
Brief Title: Study of the Efficacy of Intratumoral L19IL2 or L19TNF or L19IL2/L19TNF, in Combination with Pembrolizumab, in Unresectable Melanoma Patients
Acronym: INTACT/MeRCI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-ICKPD1-02/21; MK-3475-F20 (Other: Merck Sharp & Dohme LLC); KEYNOTE-F20 (Other: missing)
Record Dates: First submitted 2024-01-26; First posted 2024-02-29 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
MeSH Terms: conditions — Melanoma | interventions — daromun; pembrolizumab

STUDY DESIGN:
Intervention Model Description: 162 patients. Patients enrolled will be randomized in a 1:1:1 ratio. i) systemic pembrolizumab in combination with intralesional L19IL2 (Arm 1): 54 patients.
  ii) systemic pembrolizumab in combination with intralesional L19TNF (Arm 2): 54 patients iii) systemic pembrolizumab in combination with intralesional L19IL2/L19TNF (Arm 3): 54 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Systemic pembrolizumab in combination with intralesional L19IL2 (Arm 1) (Experimental): Two-weeks screening period and a 4-weeks open-label intralesional treatment period with L19IL2. Pembrolizumab will be administered by i.v. infusion on the first day of intralesional treatment with L19IL2, and will continue every 3 weeks for approximately 2 years, 35 cycles, 2 year cap or until disease progression or unacceptable toxicity, whichever comes first.
  Interventions: Drug: L19IL2; Drug: KEYTRUDA®
- Systemic pembrolizumab in combination with intralesional L19TNF (Arm 2) (Experimental): Two-weeks screening period and a 4-weeks open-label intralesional treatment period with L19TNF. Pembrolizumab will be administered by i.v. infusion on the first day of intralesional treatment with L19TNF, and will continue every 3 weeks for approximately 2 years, 35 cycles, 2 year cap or until disease progression or unacceptable toxicity, whichever comes first.
  Interventions: Drug: L19TNF; Drug: KEYTRUDA®
- Systemic pembrolizumab in combination with intralesional L19IL2/L19TNF (Arm 3) (Experimental): Two-weeks screening period and a 4-weeks open-label intralesional treatment period with L19IL2/L19TNF. Pembrolizumab will be administered by i.v. infusion on the first day of intralesional treatment with L19IL2/L19TNF, and will continue every 3 weeks for approximately 2 years, 35 cycles, 2 year cap or until disease progression or unacceptable toxicity, whichever comes first.
  Interventions: Drug: L19IL2/L19TNF; Drug: KEYTRUDA®

INTERVENTIONS:
Drug: L19IL2 — Arm 1: The amount of L19IL2 that is intratumorally administered into injectable cutaneous, subcutaneous, and nodal tumors once weekly for up to 4 weeks is dependent on the size of the tumor. The maximum dose to be administered in a single treatment visit is 13 MioIU/1 mL of L19IL2.
  Other Names: bifikafusp alfa
  Arms: Systemic pembrolizumab in combination with intralesional L19IL2 (Arm 1)
Drug: L19TNF — Arm 2: The amount of L19TNF that is intratumorally administered into injectable cutaneous, subcutaneous, and nodal tumors once weekly for up to 4 weeks is dependent on the size of the tumor. The maximum dose to be administered in a single treatment visit is 400 μg/1 mL of L19TNF.
  Other Names: onfekafusp alfa
  Arms: Systemic pembrolizumab in combination with intralesional L19TNF (Arm 2)
Drug: L19IL2/L19TNF — Arm 3: The amount of L19IL2/L19TNF that is intratumorally administered into injectable cutaneous, subcutaneous, and nodal tumors once weekly for up to 4 weeks is dependent on the size of the tumor. The maximum dose to be administered in a single treatment visit is 13MioIU L19IL2 + 400 μg L19TNF in a combined total volume of approximate 2 mL. In case that study drug-related, grade ≥ γ AEs are recorded after the first L19IL2/L19TNF dose administration, the L19TNF dose is reduced to 200 μg for the following administrations.
  Other Names: Daromun
  Arms: Systemic pembrolizumab in combination with intralesional L19IL2/L19TNF (Arm 3)
Drug: KEYTRUDA® — KEYTRUDA® will be administered by i.v. infusion as a dose of 200 mg on the first day of intralesional treatment with ICKs and will continue every 3 weeks for approximately 2 years, 35 cycles, 2 year cap or until disease progression or unacceptable toxicity, whichever comes first. ICKs intralesional treatment will be administered 30-60 minutes post administration of KEYTRUDA®.
  Other Names: pembrolizumab

SUMMARY:
The trial aims to evaluate the efficacy of single agent L19IL2, single agent L19TNF, and combination L19IL2+L19TNF given concurrently with anti-PD1 therapy compared to historical control of anti-PD-1 re-challenge alone for anti-PD1 refractory unresectable stage III-IV melanoma.

DETAILED DESCRIPTION:
The present study is a randomized, open-label, three-arm, parallel phase 2 study. A Simon two-stage design for the study of the efficacy of intralesional therapy with L19IL2 or L19TNF or L19IL2/L19TNF in combination with systemic anti-PD1 pembrolizumab immunotherapy will be used.

In the study, 162 patients will be randomized in a 1:1:1 ratio to receive:

i) systemic pembrolizumab in combination with intralesional L19IL2 (Arm 1) or ii) systemic pembrolizumab in combination with intralesional L19TNF (Arm 2) or iii) systemic pembrolizumab in combination with intralesional L19IL2/L19TNF (Arm 3).

This is an open-label study, so there is no blinding.

The study consists of a two-week screening period, followed by a 4-weeks open-label intralesional treatment period with immunocytokines (ICKs) either L19IL2, L19TNF or L19IL2/L19TNF. Pembrolizumab will be administered by i.v. infusion on the first day of intralesional treatment with ICKs, and will continue every 3 weeks for approximately 2 years, 35 cycles, 2 year cap or until disease progression or unacceptable toxicity, whichever comes first.

Follow-up for progression free survival will be performed up to 2 years after first intralesional treatment. Survival information will be collected up to 3 years after first intralesional treatment.

A safety run-in will be performed on the first 12 patients enrolled in each arm of the study. Patients will be evaluated during the first 21-days cycle for the occurrence of the treatment-related adverse events. All toxicities will be graded using NCI CTCAE Version 5.0 based on the investigator assessment to be possibly, probably, or definitely related to study treatment administration.

In addition to this, safety information collected will be routinely reviewed by the Data and Safety Monitoring Board (DSMB) in order to identify possible safety concerns.

The primary objective of the study is to demonstrate the efficacy of intralesional treatment with ICKs, in combination with systemic anti-PD1 immunotherapy with pembrolizumab, to induce objective responses in advanced melanoma patients with resistance to or progressing upon anti-PD1 checkpoint inhibitors.

Primary endpoint of the study is the Confirmed Objective Response Rate (ORR = CR + PR) in all three arms over a period of up to 2 years after first intralesional treatment, according to RECIST v1.1 criteria in each arm of the study. The primary analysis will be performed in the Intention-to-Treat population (ITT).

For each of the three treatment arms, secondary objectives include efficacy and safety of intralesional treatment with ICKs.

The secondary endpoints include:

* Best overall response (BOR; the best overall response is the best response recorded from the start of the treatment until disease progression/recurrence according to RECIST v1.1 criteria)
* Duration of response (DoR)
* Pathological response of one target lesion injected with ICKs at 18 weeks after first treatment
* Confirmed ORR over a period of up to 2 years after first intralesional treatment, according to iRECIST (see Appendix 1) and itRECIST [1] criteria in each arm of the study
* Progression-free survival (PFS) from time of randomization
* Overall survival (OS) from randomization
* Number, frequency and grading of adverse events (AEs) and serious adverse events (SAEs) related to intralesional therapy with ICKs in combination with systemic anti-PD1 therapy

End of treatment: last day of anti-PD1 therapy or until progression or unacceptable toxicity.

End of study: corresponds to the last patient last visit (LPLV).

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
2. Be > or equal to 18 years of age on day of signing informed consent.
3. Participant with histologically or cytologically confirmed diagnosis of unresectable metastatic melanoma at stage III B, C, D or IV M1a (AJCC 8th ed.). Patients with Stage IVM1b, M1c and M1d oligometastatic disease [up to 10 lesions in aggregate including lung, liver, bone or brain, with or without lymph node involvement], are eligible. However, patients with symptomatic or rapidly enlarging/bleeding brain lesions are excluded. Patients with acral lentiginous melanoma are eligible as well. Detailed information about prior therapies and burden of disease at study entry must be available.
4. Patients must have confirmed primary resistance to or acquired resistance on treatment with an anti-PD1/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria: a.) Has received at least 2 doses of an approved anti-PD-1/L1 mAb.

   b.) Has demonstrated disease progression (PD) after PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD, in the absence of rapid clinical progression. c.) Progressive disease has been documented within 12 weeks from the last dose of anti- PD-1/L1 mAb.

   i. Progressive disease is determined according to iRECIST. ii. This determination is made by the investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.
5. Patients harboring the BRAF mutation who received BRAF/MEK inhibition (or declined BRAF/MEK inhibitors) and received thereafter anti-PD1 therapy showing resistance to such immunotherapy are eligible to the study. Anti-PD1 immunotherapy must be the last therapy received by the patient prior to randomization.
6. Eligible subjects must have measurable disease (according to RECIST v1.1) as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Eligible subjects must be a candidate for intralesional therapy with at least one injectable cutaneous, subcutaneous, or nodal metastatic melanoma lesion (≥ 5 mm in longest diameter) or with multiple injectable lesions that in aggregate have a diameter of ≥ 5 mm.
7. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: a.) Not a woman of childbearing potential (WOCBP) b.) A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment. WOCBP must be using for the time period indicated highly effective contraception methods. WOCBP and effective contraception methods are defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence. Pregnancy test will be repeated at the safety visit (only WOCBP).
8. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

   Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut (details pertaining to tumor tissue submission can be found in the Procedures Manual).
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
10. Have adequate organ function as defined in the following table. Specimens must be collected within 14 days prior to the start of study treatment.
11. Be able to provide a core or excisional lymph node biopsy for biomarker analysis from an archival or newly obtained biopsy at Screening. In addition, participants may provide additional biopsy at Week 18 and at the time of discontinuation due to progression
12. Documented negative test for HIV, HBV and HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV (e.g. anti-HBsAg and/or anti-HBc Ab) a negative serum HBV-DNA test is also required.
13. All acute toxic effects (excluding alopecia and vitiligo) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v. 5.0) Grade ≤ 1 or baseline unless otherwise specified above. Note: Participants with ≤Grade β neuropathy may be eligible. Participants with endocrinerelated AEs Grade ≤β requiring treatment or hormone replacement may be eligible. Note: If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
14. Full resolution of checkpoint blockade therapy-related adverse effects (including immunerelated adverse effects) and no treatment for these AEs for at least 4 weeks prior to the time of enrollment.
15. No history of severe immune related adverse effects from prior given immune checkpoint blockade therapy (CTCAE Grade 4; CTCAE Grade 3 requiring treatment >4 weeks).
16. Male patients with WOCBP partners must agree to use simultaneously two acceptable methods of contraception (i.e. spermicidal gel plus condom) from the screening to three months following the last study drug administration. In addition, male participant must refrain from sperm donation during the treatment period.
17. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Patients with more than 10 distant melanoma lesions in lung, liver, bone or brain combined. Patients with symptomatic or rapidly enlarging/bleeding brain lesions are excluded.
2. Uveal melanoma or mucosal melanoma or melanoma with unknown primary.

   Pregnancy Exclusion
3. A WOCBP who has a positive urine pregnancy test (within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Prior/Concomitant Therapy
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher irAE.
5. Has received prior systemic anti-cancer therapy including investigational agents or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
6. Has received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis. Note: Participants must have recovered from all radiation-related toxicities and not require corticosteroids. A 1-week washout is permitted for palliative radiation (≤β weeks of radiotherapy) to non-CNS disease.
7. Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Participants who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of GVHD).
8. Has had an allogeneic tissue/solid organ transplant.
9. Has received live live or live attenuated vaccines within 30 days prior to the first dose of study treatment and while participating in the study. Note: Killed vaccines are allowed. Note: Any licensed COVID-19 vaccine (including for Emergency use) in a particular country is allowed in the study as long as they are mRNA vaccines, adenoviral vaccines, or inactivated vaccines. These vaccines will be treated just as any other concomitant therapy. Investigational vaccines (i.e., those not licensed or approved for Emergency Use) are not allowed.

   Diagnostic assessments
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
11. Has a known additional malignancy that is progressing or has required active treatment within the past two (2) years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder tumors (Ta, Tis & T1), second primary melanoma in situ, or carcinoma in situ, that have undergone potentially curative therapy are not excluded.
12. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
13. Has severe hypersensitivity (≥Grade γ) to pembrolizumab and/or any of its excipients, or to (immuno)cytokines IL2, TNF and/or any of its excipients
14. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

    Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
15. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
16. Has an active infection requiring systemic therapy.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
18. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
19. Previous enrolment and randomization in this same study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) | Evaluated over a period of up to 2 years after first intralesional treatment. TA visits will be performed at week 12, 18, 24, 36, 48, 64, 80 and 96 after first intralesional treatment or until confirmed progression or death, whichever occurs first
  Objective Response Rate (ORR = CR + PR) in all three arms to demonstrate the efficacy of intralesional treatment with immunocytokines (L19IL2, or L19TNF, or L19IL2/L19TNF), in combination with the systemic anti-PD1 pembrolizumab, to induce objective responses in advanced melanoma patients with resistance to or progressing upon anti-PD1 checkpoint inhibitors. The primary analysis will be performed in the Intention-to-Treat population (ITT).
  Assessed during Tumor Assessment (TA) visits.

SECONDARY OUTCOMES:
Best overall response (BOR) | From the date of first treatment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 96 Weeks
  Best response recorded from the start of the treatment until disease progression/recurrence after first treatment according to RECIST v1.1 criteria
Duration of Response (DoR) | From the date of first treatment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 36 Months
  Time from first documented evidence of CR or PR until first documented disease progression or death due to any cause. DoR will be summarized descriptively using Kaplan-Meier medians and quartiles.
Pathological response | At 18 weeks after first treatment
  Histopathological analysis will be performed on biopsies obtained at baseline and at Week 18 for one target injected lesions.
  This is to determine:
  * Confirmation of melanoma metastasis( Biopsy at baseline)
  * Presence of residual tumor cells (%, biopsy at week 18),
  * Presence of Necrosis % (biopsy at week 18),
  * Presence of melanosis/fibrosis % (biopsy at weeks 18 after first treatment)
Confirmed ORR | From date of first administration, after a period of up to 2 years
  Confirmed ORR over a period of up to 2 years after first intralesional treatment according to iRECIST and itRECIST criteria in each arm of the study
Progression-free survival (PFS) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 96 Weeks
  Difference between date of randomization and the date of progression according to RECIST v. 1.1 criteria or death
Overall survival (OS) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 96 Weeks
  Difference between date of randomization and the date of death for any cause
Serious Adverse Event (SAEs) | From date of ICF signature until first follow-up visit (Week 12). Subsequently only AEs and SAEs (and related medications or procedures) that were judged as drug or study related will be recorded, up to week 96
  Percentage of Patients in Each Treatment Group with Drug-Related Adverse Events, Serious Adverse Event (SAEs)
Drug-Induced Liver Injury (DILI) | From date of ICF signature until first follow-up visit (Week 12). Subsequently only DILI that were judged as drug or study related will be recorded, up to week 96
  Number of patients with Drug-Induced Liver Injury (DILI)
Number of patients with Adverse Events of Special Interest (AESI) | From date of ICF signature until first follow-up visit (Week 12). Subsequently only AESI that were judged as drug or study related will be recorded, up to week 96
Number of patients with Immune-Related Adverse Events (IRAEs) | From date of ICF signature until first follow-up visit (Week 12). Subsequently only IRAEs that were judged as drug or study related will be recorded, up to week 96
Number of participants with abnormal hematology laboratory tests results | From the screening to the last visit (Week 103)
  Red Blood cells; Millions/microliter (M/mcL)
Number of participants with abnormal hematology laboratory tests results | From the screening to the last visit (Week 103)
  Count of absolute neutrophil (ANC), White Blood cells (WBC), Platelet, Differential; thousands/microliter (K/mcL)
Number of participants with abnormal hematology laboratory tests results | From the screening to the last visit (Week 103)
  Hematocrit; percent (%)
Number of participants with abnormal hematology laboratory tests results | From the screening to the last visit (Week 103)
  Hemoglobin; grams/deciliter (g/dL)
Number of participants with abnormal serum chemistry laboratory tests results | From the screening to the last visit (Week 103)
  Creatinine, Blood Urea Nitrogen or Urea, Uric acid, Calcium, Glucose, Phosphorus, Magnesium; milligrams/deciliter (mg/dL)
Number of participants with abnormal serum chemistry laboratory tests results | From the screening to the last visit (Week 103)
  Potassium, Sodium, Chloride; milliequivalents/liter (mEq/L)
Number of participants with abnormal serum chemistry laboratory tests results | From the screening to the last visit (Week 103)
  Total proteins, Albumin; grams/deciliter (g/dL)
Number of participants with abnormal serum chemistry laboratory tests results | From the screening to the last visit (Week 103)
  Lactate dehydrogenase (LDH); units/liter (U/L)
Number of participants with abnormal serum chemistry laboratory tests results | From the screening to the last visit (Week 103)
  Adrenocorticotropic Hormone (ACTH); picograms/milliliter (pg/ml)
Number of participants with abnormal coagulation laboratory tests results | From the screening to the last visit (Week 103)
  Prothrombin Time PT or PT INR, PTT or aPTT; seconds (sec)
Number of participants with abnormal body temperature | From the screening to the last visit (Week 103)
  Body temperature; degree centigrade
Number of participants with abnormal blood pressure | From the screening to the last visit (Week 103)
  Systolic and diastolic blood pressure (after 3 minutes in sitting position); mmHg
Number of participants with abnormal Electrocardiogram (ECG) readings | At the screening visit, at Visit 6 (week 5) and at Visit 12 (week 18)
  Heart rate, standard intervals (PR, QRS, QT, and QTc) and any observed abnormality; millisecond
Number of participants with abnormal Echocardiogram (ECHO) readings | At the screening visit, at Visit 6 (week 5) and at Visit 12 (week 18)
  Morphological and functional aspects of the heart. Left Ejection Fraction (LVEF) is determined; percentage %
Number of participants with abnormal physical examination results | From the screening to first follow up visit
Concomitant medication usage | From the screening and throughout study
Assessment of the formation of human anti-fusion protein antibodies (HAFA) against L19IL2 and L19TNF | At weeks 1, 2 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Bello, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States